CLINICAL TRIAL: NCT04621292
Title: Prospective Comparative Study of the SoCoLoc vs ISAR Scales for the Identification of Complex Elderly Patients in the Emergency Department of the Annecy Genevois Hospital.
Brief Title: Prospective Study Assessing Two Scales for Identification of Complex Elderly Patients in the Emergency Department
Acronym: SOCOLOC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Annecy Genevois (Other)
Responsible Party: Sponsor
Other Study IDs: 20-05
Record Dates: First submitted 2020-11-03; First posted 2020-11-09 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Geriatric

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
With the help of medical progress, life expectancy has increased in our country, resulting in an increase in the number of elderly people and especially so-called complex patients. These complex elderly patients present with a combination of poly pathology, locomotor disorders and loss of autonomy, which leads to increased risks of hospitalization, re-hospitalization or difficulty in remaining at home. These risks could be reduced by early adapted care specific to this type of patient. To do this, it is necessary to identify these complex elderly patients as early as possible in their care pathway.

Screening complex elderly patients in the emergency department would require trained and educated staff, or the use of a simple, rapid and reliable diagnostic scale. The purpose of this study is to compare two scales for the screening of complex elderly patients, whose use is adapted to the Hospital Emergency Department environment.

This study assess the diagnostic performance of the ISAR and SoCoLoc scales for complex elderly patients.

DETAILED DESCRIPTION:
The assumption of the study is that at least one of these two scales (ISAR or SoCoLoc) is adapted to the constraints of hospital emergencies and that it presents good performances for the screening of elderly patients in complex medico-social situations (sensitivity ≥ 90% and specificity ≥ 50%).

ELIGIBILITY:
Inclusion Criteria:

* Patients over 75 years of age
* Patient presenting to the "Emergency Department" of the Annecy Genevois hospital, whatever the reason for consultation, from Monday to Friday between 8:00 a.m. and 8:00 p.m.
* Patient informed of the study and not opposed to participation

Exclusion Criteria:

* Patients under guardianship or curatorship
* Patients under the safeguard of justice
* Patient presenting for a life-threatening emergency
* Patient unable to answer the questions on the scales
* Patient does not speak French
* Patients who have already been included in the study: any patient already included in the study and making another trip to the emergency department cannot be included a second time.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: The study will focus on patients aged 75 and over who consult the Emergency Department of the Annecy Geneva Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2020-08-17 (Actual); Primary Completion 2020-10-16 (Actual); Study Completion 2020-10-16 (Actual)

PRIMARY OUTCOMES:
Overall diagnostic performance of the two scales comparing the AUC | Up to emergency admission
  The overall diagnostic performance of each scale will be measured using the area under the ROC curve (sensitivity vs. 1-specificity).
  The performance of the two scales will be measured and compared using a parametric or non-parametric Z-test for matched data according to the number of events observed, i.e. the number of "complex" patients. A ROC curve will be performed in order to determine the best positivity threshold of each scale.
  Patients will be classified as "complex" or "non-complex" by the blind adjudication committee of the results of the two scales.

SECONDARY OUTCOMES:
Sensitivity and specificity of the two scales | Up to emergency admission
  Sensitivity, specificity, positive predictive value, negative predictive value, positive likelihood ratio and negative likelihood ratio of SoCoLoc and ISAR
Number and proportion of complex elderly patients | Up to emergency admission
  Number and proportion of complex elderly patients, as well as its 95% confidence interval, evaluated according to the definition accepted by the adjudication committee.
Patient characteristics description | Up to emergency admission
  Description of patient characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Bahman MOHEB KHOSRAVI, Principal Investigator — CH Annecy Genevois
Locations (1):
- Centre Hospitalier Annecy Genevois, Metz-Tessy, France